CLINICAL TRIAL: NCT01259713
Title: A Phase 3, Double-Blind, Multicenter, Randomized, Placebo-Controlled Study to Assess the Efficacy, Safety and Tolerability of Prophylactic Liposomal Amphotericin B (AmBisome®) for the Prevention of Invasive Fungal Infections (IFIs) in Subjects Receiving Remission-Induction Chemotherapy for Acute Lymphoblastic Leukemia (ALL)
Brief Title: Prevention of Invasive Fungal Infections (IFIs) in Subjects Receiving Chemotherapy for Acute Lymphoblastic Leukemia
Acronym: AmBiGuard
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GS-EU-131-0247; 2010-019562-91 (EudraCT Number)
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Invasive Fungal Disease
Keywords: Ambisome; ALL; invasive fungal infection; prophylaxis; liposomal amphotericin B; Invasive fungal infection prophylaxis
MeSH Terms: conditions — Invasive Fungal Infections | interventions — liposomal amphotericin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal amphotericin B (Experimental): Liposomal amphotericin B 5 mg/kg twice weekly administered by IV route over 2 hours twice weekly (each dose separated alternately by 2 and 3 days each week) during induction chemotherapy
  Interventions: Drug: Liposomal amphotericin B
- Placebo (Placebo Comparator): Placebo to match liposomal amphotericin B twice weekly administered by IV route over 2 hours twice weekly (each dose separated alternately by 2 and 3 days each week) during induction chemotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liposomal amphotericin B — Ambisome 5 mg/kg twice weekly administered by IV route over 2 hours twice weekly (each dose separated alternately by 2 and 3 days each week during induction chemotherapy
  Other Names: AmBisome
  Arms: Liposomal amphotericin B
Drug: Placebo — Placebo to match liposomal amphotericin B administered by IV route over 2 hours twice weekly (each dose separated alternately by 2 and 3 days each week) during induction chemotherapy
  Arms: Placebo

SUMMARY:
The study aims to investigate whether prophylaxis with liposomal amphotericin B (AmBisome®) can reduce the incidence of invasive fungal infections (IFIs) in patients with Acute Lymphoblastic Leukemia (ALL) who are undergoing their first remission induction.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ALL receiving an ALL chemotherapy regimen that typically induces at least 10 days of neutropenia defined as an absolute neutrophil count < 500 cells/mm^3 or 0.5 × 10^9 cells/L

  * Subjects with lymphoblastic lymphoma or any malignancy other than ALL are NOT eligible for this study.
* Age ≥ 18 years
* Able to have all screening tests performed quickly to ensure results can be obtained and evaluated before randomization so that the first dose of randomized study drug for IFI prophylaxis can be administered within 5 days of first remission-induction chemotherapy

  * Preremission induction treatment (ie, pre-phase) with a minimally or nonmyelosuppressive regimen for up to one week is not considered to constitute the beginning of remission induction chemotherapy
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures

Exclusion Criteria:

* Known hypersensitivity to amphotericin B or AmBisome, the metabolites or formulation excipients, in particular known history of anaphylactic reaction to amphotericin B or AmBisome or any of its metabolites or formulation excipients
* Known hypersensitivity to the excipients of the placebo formulation
* Current fever (≥ 38°C) unless explained by noninfectious causes
* Subjects with proven, probable or possible IFI (according to European Organization for the Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG) criteria) at screening or in subject history
* Pulmonary infiltrates
* Concomitant or previous treatment with an antifungal drug within the previous 30 days unless the plasma level is below the limit of detection or at least 5 half-lives of the antifungal has elapsed since the treatment was given
* Serum creatinine > 2 × the upper limit of the normal range (ULN)
* Grade 3 Liver function test results: alanine aminotransferase or aspartate aminotransferase > 5 × ULN; total bilirubin > 2.5 x ULN
* Any severe co morbidity other than underlying hematological disease (ALL), which in the investigator's judgment may interfere with study evaluations or affect the subject's safety
* Subjects who have taken any investigational drug in the last 30 days prior to screening, with the exception of ALL chemotherapy investigational products being used as part of the subject's current ALL treatment protocol
* Pregnant or nursing females
* Subjects with a prior history of a malignancy that was treated with a myeloablative chemotherapy regimen are NOT eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Hawkins, MD, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 86 study sites. The first participant was screened on 13 April 2011. The last study visit occurred on 29 January 2014.
Pre-assignment Details: 391 participants were screened.
Groups:
- Liposomal Amphotericin B: Liposomal amphotericin B (AmBisome®) 5 mg/kg twice weekly administered by IV route over 2 hours twice weekly (each dose separated alternately by 2 and 3 days each week) during induction chemotherapy
Period: Overall Study
Arm/Group | Liposomal Amphotericin B | Placebo
Started | 237 | 118
Completed | 142 | 77
Not Completed | 95 | 41
Not completed — Adverse Event | 54 | 23
Not completed — Death Not Related to IFI | 8 | 1
Not completed — Investigators Discretion | 14 | 6
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 5 | 4
Not completed — Subject Withdrew Consent | 12 | 7

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Amphotericin B | Placebo | Total
Number analyzed (Participants) | 237 | 118 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (15.16) | 44.8 (17.52) | 44.6 (15.96)
Age, Customized [Number; unit: participants]
  ≤ 25 years | 37 | 25 | 62
  > 25 to ≤ 60 years | 160 | 64 | 224
  > 60 years | 40 | 29 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 58 | 156
  Male | 139 | 60 | 199
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black | 4 | 3 | 7
  White | 211 | 100 | 311
  Not Permitted | 17 | 15 | 32
  Other | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Germany | 52 | 23 | 75
  Italy | 41 | 25 | 66
  France | 33 | 19 | 52
  Belgium | 20 | 11 | 31
  Spain | 21 | 7 | 28
  Greece | 14 | 13 | 27
  Portugal | 13 | 4 | 17
  Turkey | 7 | 4 | 11
  Austria | 6 | 3 | 9
  Israel | 9 | 0 | 9
  Switzerland | 6 | 1 | 7
  Brazil | 8 | 7 | 15
  Argentina | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Proven or Probable IFIs During Remission-induction Chemotherapy for Acute Lymphoblastic Leukemia (ALL)
Description: Diagnoses of proven or probable invasive fungal infections (IFI) were assessed according to European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG) criteria by the independent data review board (IDRB) who were blinded to treatment assignment.
  The duration of remission-induction chemotherapy was defined as the period from the initiation of remission-induction chemotherapy administration to the start of consolidation or salvage therapy.
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: Intent-to-Treat (ITT) Analysis Set: participants in the safety analysis set who had no major violations of entrance criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
percentage of participants | 7.9 | 11.7
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; A two-group Cochran-Mantel-Haenszel (CMH) test with a 0.05 two-sided significance level and 2:1 allocation of 354 randomized subjects (236 AmBisome, 118 placebo) would have 81% power to detect a relative reduction of 75% if the rate of IFI is 10% in the placebo group (based on unpublished data from the German Multicenter Acute Lymphoblastic Leukemia Working Group (GMALL) and consistent with the published rate of 16.4% in patients with hematological malignancies undergoing remission induction); Test type: Non-Inferiority or Equivalence — For the interim analysis performed when 50% of the subjects had completed the study, an alpha of 0.0003 was spent. Therefore, the significance level for the 2-sided test in the primary analysis at the end of the study was 0.0497 (corresponding to 95.03% confidence interval (CI)); p = 0.24, Cochran-Mantel-Haenszel — P-value was from a stratum-adjusted (stratified by region) CMH test; Relative risk reduction = 0.33, 95.03% CI 2-sided [-0.32 to 0.66] — Relative risk reduction = 1 - risk ratio

2. Secondary Outcome: Percentage of Participants With Pulmonary Infiltrates According to the Central Image Reader
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
percentage of participants | 20.2 | 27.0
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Test type: Superiority or Other; p = 0.15, Cochran-Mantel-Haenszel — P-value was from a stratum-adjusted (stratified by region) CMH test; Relative risk reduction = 0.25, 95% CI 2-sided [-0.11 to 0.50] — Relative risk reduction = 1 - risk ratio

3. Secondary Outcome: Percentage of Participants Diagnosed With Proven or Probable IFIs According to the EORTC/MSG Criteria, as Assessed by the Investigator
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
percentage of participants | 11.0 | 10.8
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Test type: Superiority or Other; p = 0.97, Cochran-Mantel-Haenszel — P-value was from a stratum-adjusted (stratified by region) CMH test; Relative risk reduction = -0.01, 95% CI 2-sided [-0.94 to 0.47] — Relative risk reduction = 1 - risk ratio

4. Secondary Outcome: Time to Diagnosis of Proven or Probable IFIs According to the EORTC/MSG Criteria, as Assessed by the IDRB.
Description: Time to diagnosis of proven or probable IFIs is presented as the median (Q1,Q3) days to diagnosis of those participants who experienced a proven or probable IFI. Median was not reached if < 50% of participants had an event; Q1 was not reached if < 25% of participants had an event; Q3 was not reached if < 75% of participants had an event.
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
days | NA [NA to NA] — NA = Not reached | NA [NA to NA] — NA = Not reached
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Test type: Superiority or Other; p = 0.33, Log Rank — The p-value is from the log-rank test stratified by region

5. Secondary Outcome: Percentage of Participants Requiring Antifungal Treatment During Remission-Induction Chemotherapy
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
percentage of participants | 16.2 | 21.6
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Test type: Superiority or Other; p = 0.22, Cochran-Mantel-Haenszel — P-value was from a stratum-adjusted (stratified by region) CMH test; Relative risk reduction = 0.25, 95% CI 2-sided [-0.19 to 0.53] — Relative risk reduction = 1 - risk ratio

6. Secondary Outcome: Percentage of Participants Who Died Due to Fungal Infection; Causality as Assessed by the IDRB.
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
percentage of participants | 0.9 | 0
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Test type: Superiority or Other; p = 0.32, Cochran-Mantel-Haenszel — P-value was from a stratum-adjusted (stratified by region) CMH test

7. Secondary Outcome: Percentage of Participants Who Died Due to Fungal Infection; Causality as Assessed by the Investigator.
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
percentage of participants | 0.9 | 0
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Test type: Superiority or Other; p = 0.32, Cochran-Mantel-Haenszel — P-value was from a stratum-adjusted (stratified by region) CMH test

8. Secondary Outcome: Time From Beginning of Remission-induction Chemotherapy Until the Beginning of Consolidation Therapy
Description: This endpoint was to evaluate the potential impact of IFI prevention on the efficacy of remission-induction chemotherapy for ALL.
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
days | 50 [38 to 75] | 55 [36 to 75]
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Test type: Superiority or Other; p = 0.69, Log Rank — The p-value was from the log-rank test stratified by region; Participants without consolidation/salvage therapy dates were censored using the earlier of the Early Termination and Study Completion dates

9. Secondary Outcome: Percentage of Participants With Complete Remission at the End of Remission Induction
Description: as for outcome 8
Time Frame: During remission-induction chemotherapy (average 7 weeks)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Amphotericin B | Placebo
Number analyzed (Participants) | 228 | 111
percentage of participants | 72.8 | 79.3
Statistical Analysis 1: Comparison: Liposomal Amphotericin B vs Placebo; Participants were not stratified for leukemia risk; Test type: Superiority or Other; p = 0.20, Cochran-Mantel-Haenszel — P-value was from a stratum-adjusted (stratified by region) CMH test; Relative risk reduction = 0.08, 95% CI 2-sided [-0.04 to 0.19] — Relative risk reduction = 1 - risk ratio

ADVERSE EVENTS:
Time Frame: From first dose to last dose of study drug plus 30 days.
Description: Safety Analysis Set; participants who were randomized and received at least 1 dose of study drug.
  The duration of remission-induction chemotherapy was defined as the period from the initiation of remission-induction chemotherapy administration to the start of consolidation or salvage therapy.
Arm/Group | Liposomal Amphotericin B | Placebo
Serious Adverse Events (participants affected / at risk) | 79/237 | 38/118
Other Adverse Events (participants affected / at risk) | 233/237 | 114/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Amphotericin B (N=237) | Placebo (N=118)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 4 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0
Ileitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Systemic inflammatory response syndrome (General disorders) | 0 | 2
Chestpain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Allergic oedema (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Septic shock (Infections and infestations) | 13 | 2
Pneumonia (Infections and infestations) | 7 | 3
Sepsis (Infections and infestations) | 4 | 6
Device related infection (Infections and infestations) | 3 | 0
Bacterial sepsis (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pseudomonal sepsis (Infections and infestations) | 2 | 0
Aspergillus infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1
Respiratory moniliasis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Blood creatinine increased (Investigations) | 3 | 0
Creatinine renal clearance decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 2
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0
Meningism (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 2
Renal failure acute (Renal and urinary disorders) | 3 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Amphotericin B (N=237) | Placebo (N=118)
Anaemia (Blood and lymphatic system disorders) | 49 | 27
Febrile neutropenia (Blood and lymphatic system disorders) | 50 | 26
Neutropenia (Blood and lymphatic system disorders) | 40 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 42 | 14
Coagulopathy (Blood and lymphatic system disorders) | 13 | 9
Tachycardia (Cardiac disorders) | 13 | 8
Vertigo (Ear and labyrinth disorders) | 14 | 8
Nausea (Gastrointestinal disorders) | 118 | 50
Vomiting (Gastrointestinal disorders) | 75 | 43
Constipation (Gastrointestinal disorders) | 74 | 40
Diarrhoea (Gastrointestinal disorders) | 66 | 36
Abdominal pain (Gastrointestinal disorders) | 55 | 35
Abdominal pain upper (Gastrointestinal disorders) | 39 | 14
Haemorrhoids (Gastrointestinal disorders) | 18 | 12
Stomatitis (Gastrointestinal disorders) | 14 | 11
Dyspepsia (Gastrointestinal disorders) | 14 | 4
Pyrexia (General disorders) | 65 | 37
Mucosal inflammation (General disorders) | 61 | 32
Oedema peripheral (General disorders) | 56 | 18
Asthenia (General disorders) | 32 | 19
Fatigue (General disorders) | 17 | 10
Chest pain (General disorders) | 18 | 8
Chills (General disorders) | 17 | 9
Oedema (General disorders) | 15 | 6
Pain (General disorders) | 10 | 11
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 7
Oral herpes (Infections and infestations) | 22 | 7
Oral candidiasis (Infections and infestations) | 8 | 11
Bacterial infection (Infections and infestations) | 12 | 6
Pneumonia (Infections and infestations) | 15 | 3
Folliculitis (Infections and infestations) | 10 | 6
Antithrombin III decreased (Investigations) | 33 | 14
Blood fibrinogen decreased (Investigations) | 19 | 8
Alanine aminotransferase increased (Investigations) | 17 | 9
Aspartate aminotransferase increased (Investigations) | 19 | 4
Blood bilirubin increased (Investigations) | 16 | 4
Blood creatinine increased (Investigations) | 20 | 0
Weight decreased (Investigations) | 13 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 83 | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 24 | 9
Decreased appetite (Metabolism and nutrition disorders) | 18 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 18 | 7
Fluid retention (Metabolism and nutrition disorders) | 15 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 13 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 14 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Headache (Nervous system disorders) | 84 | 45
Dizziness (Nervous system disorders) | 11 | 12
Paraesthesia (Nervous system disorders) | 14 | 9
Insomnia (Psychiatric disorders) | 32 | 17
Anxiety (Psychiatric disorders) | 19 | 15
Depression (Psychiatric disorders) | 12 | 5
Agitation (Psychiatric disorders) | 5 | 7
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Rash (Skin and subcutaneous tissue disorders) | 39 | 11
Erythema (Skin and subcutaneous tissue disorders) | 19 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 4
Hypotension (Vascular disorders) | 17 | 15
Hypertension (Vascular disorders) | 12 | 7
Haematoma (Vascular disorders) | 15 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years